CLINICAL TRIAL: NCT05617495
Title: Targeting Adolescent Depression Symptoms Using Network-based Real-time fMRI Neurofeedback and Mindfulness Meditation (NIMH); Mindfulness-Based Real-Time fMRI Neurofeedback for Depression (IRB)
Brief Title: Mindfulness-Based fMRI Neurofeedback for Depression
Acronym: mbNF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Randy P. Auerbach, Ph.D., ABPP, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAV1161; R61MH132072-01 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Depression in Adolescence; Rumination
Keywords: Real-time fMRI Neurofeedback; Mindfulness; Rumination; Major Depressive Disorder
MeSH Terms: conditions — Rumination Syndrome; Depressive Disorder, Major | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 15-Minute mbNF (Active Comparator): Participants receiving mindfulness training and 15-minute session of mbNF
  Interventions: Other: Mindfulness + fMRI Neurofeedback
- 30-Minute mbNF (Active Comparator): Participants receiving mindfulness training and 30-minute session of mbNF
  Interventions: Other: Mindfulness + fMRI Neurofeedback

INTERVENTIONS:
Other: Mindfulness + fMRI Neurofeedback — Prior to neurofeedback, participants will receive 45 minutes of mindfulness training. Participants will then receive mindfulness-based fMRI neurofeedback targeting the default mode network and frontoparietal control network.
  Other Names: Mindfulness-based Real-time fMRI Neurofeedback

SUMMARY:
In the United States, adolescents experience alarmingly high rates of major depression, and gold-standard treatments are only effective for approximately half of patients. Rumination may be a promising treatment target, as it is well-characterized at the neural level and contributes to depression onset, maintenance, and recurrence as well as predicts treatment non-response. Accordingly, the proposed research will investigate whether an innovative mindfulness-based real-time functional magnetic resonance imaging (fMRI) neurofeedback intervention successfully elicits change in the brain circuit underlying rumination to improve clinical outcomes among depressed adolescents.

DETAILED DESCRIPTION:
Adolescent major depressive disorder (MDD) is common and debilitating. Presently, gold-standard treatments are only effective for approximately half of patients, underscoring the need to develop novel interventions, particularly to target core underlying mechanisms and more effectively treat this recurrent disorder.

Rumination, the tendency to perseverate about depressive symptoms, contributes to MDD onset and predicts treatment non-response and relapse. At the neural level, rumination is characterized by elevated functional connectivity within the default mode network (DMN), and similarly, prior research has consistently demonstrated patterns of DMN hyper-connectivity in MDD. Interestingly, mindfulness meditation, which trains attentional focus to the present moment, reduces perseverative thinking, ruminative tendencies, and depression symptoms. Further, our research and others have shown that adolescents can apply mindfulness practices to decrease perceived stress, increase sustained attention, and suppress DMN activity. Although mindfulness has profound mental health benefits, for some, mindfulness alone may not be sufficient to mitigate ruminative tendencies during a depressive episode. That is, MDD symptoms, including reduced motivation, inattention, and lack of self-efficacy, may impede a patient's progress in successfully acquiring and utilizing mindfulness strategies necessary to change perceptions about one's environment and relationships. To directly address this challenge, this project will use real-time fMRI neurofeedback to enhance the acquisition and utilization of mindfulness skills to better target DMN hyper-connectivity, rumination, and depressive symptoms.

Specifically, a novel, mindfulness-based, real-time neurofeedback (mbNF) paradigm will be used whereby people observe a visual display of their brain activity and practice mindfulness to volitionally reduce DMN activation. Adolescents (N=90; ages 13-18 years) diagnosed with MDD will complete a ~45-minute mindfulness training outside the MRI scanner. To test target engagement of reducing DMN hyper-connectivity and dosing effects, adolescents will all receive mbNF and changes in brain connectivity will be examined (primary outcome). To examine dosing effects, adolescents will be randomized to receive either a 15- or a 30-minute mbNF session (n=45/dose group). Clinician-administered instruments, self-reports, and smartphone ecological momentary assessment will be used test whether mbNF contributes to a greater reduction in clinician assessed depression symptoms as well as decreased rumination post-treatment (secondary outcomes). As a whole, mbNF is directly in line with precision medicine initiatives, and if successful, could revolutionize clinical care for depressed adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-18 years-old
* Written informed assent/consent and parental/guardian permission for 13-17 year-olds or informed consent for 18 year-olds
* Tanner puberty stage ≥3
* Meets current diagnostic criteria for MDD
* English fluency

Exclusion Criteria:

* Lifetime history of primary psychotic disorders, bipolar disorder, oppositional defiant disorder, conduct disorder, developmental disorder (e.g., autism), post-traumatic stress disorder, or eating disorders
* Substance use disorder, moderate or severe in past 6 months
* Active suicidal ideation with a specific plan
* History of seizure disorder
* Medical or neurological illness (e.g., severe head injury)
* MRI contraindications
* Current psychotropic medication use other than antidepressant medication
* Intelligence quotient (IQ) <80.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Within-person Default Mode Network (DMN) Connectivity | Pre-mbNF procedure
  DMN change will be assessed via fMRI from before mbNF.
Within-person Default Mode Network (DMN) Connectivity | Post-mbNF procedure
  DMN connectivity will be assessed via fMRI from post mbNF. Changes in DMN connectivity following mbNF are anticipated.

SECONDARY OUTCOMES:
Self-Report Depression Symptoms | Pre-mbNF procedure
  Self-report of depression symptoms from pre-mbNF assessed through the Mood and Feelings Questionnaire; 33-items with each item ranging from 0-2; Higher scores reflect greater depression
Self-Report Depression Symptoms | Immediately Post-mbNF procedure
  Self-report of depression symptoms from post-mbNF assessed through the Mood and Feelings Questionnaire; 33-items with each item ranging from 0-2; Higher scores reflect greater depression
Self-Report Depression Symptoms | 1-month
  Self-report of depression symptoms from 1 month after mbNF assessed through the Mood and Feelings Questionnaire; 33-items with each item ranging from 0-2; Higher scores reflect greater depression
Interviewer-Assessed Depression Symptoms | Baseline
  Depressive symptoms at baseline assessed via the Children's Depression Rating Scale - Revised, which is a clinician interview of depression symptoms. Scores range from 17 to 119 with higher scores reflecting greater depression symptom severity.
Interviewer-Assessed Depression Symptoms | 1-month
  Depressive symptoms at 1-month post mbNF assessed via the Children's Depression Rating Scale - Revised, which is a clinician interview of depression symptoms. Scores range from 17 to 119 with higher scores reflecting greater depression symptom severity.
Self-Reported Rumination | Immediately Post-mbNF procedure
  Self-report of rumination symptoms pre-mbNF assessed through the Ruminative Response Scale; 22-items with each item ranging from 1-4; Higher scores reflect greater rumination
Self-Reported Rumination | Immediately Post-mbNF procedure
  Self-report of rumination symptoms from post-mbNF assessed through the Ruminative Response Scale; 22-items with each item ranging from 1-4; Higher scores reflect greater rumination
Self-Reported Rumination | 1-month
  self-report of rumination symptoms 1-month post mbNF assessed through the Ruminative Response Scale; 22-items with each item ranging from 1-4; Higher scores reflect greater rumination

OTHER OUTCOMES:
Ecological Momentary Assessment of Depression Symptoms | Immediately Post-mbNF procedure
  Change in self-report of depressive symptoms from baseline to post-mbNF assessed through the Patient Health Questionnaire (PHQ)-2 delivered via ecological momentary assessment over a 7-day period; 2-items with each item ranging from 0-100; Higher scores reflect greater depression severity.
Ecological Momentary Assessment of Depression Symptoms | 1-month
  Change in self-report of depressive symptoms from baseline to 1-month post-mbNF assessed through the Patient Health Questionnaire (PHQ)-2 delivered via ecological momentary assessment over a 7-day period; 2-items with each item ranging from 0-100; Higher scores reflect greater depression severity.
Ecological Momentary Assessment of Rumination | Immediately Post-mbNF procedure
  Change in self-report of rumination (5-items) from baseline to post-mbNF assessed via ecological momentary assessment over a 7-day period; 5-items with each item ranging from 0-100; Higher scores reflect greater rumination.
Ecological Momentary Assessment of Rumination | 1-month
  Change in self-report of rumination (5-items) from baseline to 1-month post-mbNF assessed via ecological momentary assessment over a 7-day period; 5-items with each item ranging from 0-100; Higher scores reflect greater rumination.
Ecological Momentary Assessment of Mindfulness | Immediately Post-mbNF procedure
  Change in self-report of mindfulness (3-items) from baseline to post-mbNF assessed via ecological momentary assessment over a 7-day period; 3-items with each item ranging from 0-100; Higher scores reflect greater mindfulness.
Ecological Momentary Assessment of Mindfulness | 1-month
  Change in self-report of mindfulness (3-items) from baseline to 1-month post-mbNF assessed via ecological momentary assessment over a 7-day period; 3-items with each item ranging from 0-100; Higher scores reflect greater mindfulness.
Default Mode Network (DMN) and Frontoparietal Control Network (FPCN) Connectivity | Immediately Post-mbNF procedure
  Anticorrelation between DMN and FPCN will be assessed via fMRI from pre and post mbNF. Changes in DMN-FPCN anticorrelation are anticipated.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northeastern University, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
We will upload de-identified data to the NIMH NDA.

REFERENCES:
- [Derived] Bloom PA, Pagliaccio D, Zhang J, Bauer CCC, Kyler M, Greene KD, Treves I, Morfini F, Durham K, Cherner R, Bajwa Z, Wool E, Olafsson V, Lee RF, Bidmead F, Cardona J, Kirshenbaum JS, Ghosh S, Hinds O, Wighton P, Galfalvy H, Simpson HB, Whitfield-Gabrieli S, Auerbach RP. Mindfulness-based real-time fMRI neurofeedback: a randomized controlled trial to optimize dosing for depressed adolescents. BMC Psychiatry. 2023 Oct 17;23(1):757. doi: 10.1186/s12888-023-05223-8. PMID 37848857